CLINICAL TRIAL: NCT02745015
Title: Effect of Non Surgical Treatment of Periodontitis on Glycaemic Control in a Type 2 Diabetic Populations of Cameroon
Brief Title: Effect of Non Surgical Treatment of Periodontitis on Diabetes Control
Acronym: PARODIA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, Sobngwi Eugene, Professor, Yaounde Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNO20154
Record Dates: First submitted 2016-04-16; First posted 2016-04-20 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Periodontitis; Diabetes
Keywords: periodontitis; diabetes; HbA1c; inflammation
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Experimental): immediate non-surgical periodontal treatment
  Interventions: Procedure: non-surgical periodontal treatment
- control (Other): non-surgical periodontal treatment scheduled for the following 3-monthly visit
  Interventions: Procedure: non-surgical periodontal treatment

INTERVENTIONS:
Procedure: non-surgical periodontal treatment — full-mouth scaling and root planing

SUMMARY:
The aim of this study is to investigate the effects of non-surgical periodontal treatment on the metabolic control of type2 diabetes patients. Patients with type two diabetes mellitus patients and confirmed chronic periodontitis will be selected and randomly assign to two groups. The treatment group will receive immediate full-mouth scaling and root planing whereas the control group will be scheduled to receive periodontal treatment at the following 3-month visit. Plaque index, bleeding index, probing pocket depth, recessions and cervical attachment loss will be recorded at baseline, at six weeks and at three months. Glycated haemoglobin (HbA1c) and C-reactive protein (CRP) will be analysed at baseline and three months following enrolment.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of non-surgical periodontal treatment on the metabolic control of type2 diabetes patients. Patients with type two diabetes mellitus patients and confirmed chronic periodontitis will be selected and randomly assign to two groups. The treatment group will receive immediate full-mouth scaling and root planing whereas the control group will be scheduled to receive periodontal treatment at the following 3-month visit. Plaque index, bleeding index, probing pocket depth, recessions and cervical attachment loss will be recorded at baseline, at six weeks and at three months. Glycated haemoglobin (HbA1c) and C-reactive protein (CRP) will be analysed at baseline and three months following enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least one year
* periodontitis
* HbA1c > 7%

Exclusion Criteria:

* Periodontal treatment in the last 6 months
* antibiotics in the last 3 months
* tobacco smoking
* pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Metabolic | 3 months
  Change in HbA1c

SECONDARY OUTCOMES:
Inflammation | 3 months
  change in CRP level between baseline and 3-month post intervention
Periodontal 1 | 3 months
  Change in plaque index between baseline and 3-month post intervention
Periodontal 2 | 3 months
  Change in bleeding index between baseline and 3-month post intervention
Periodontal 3 | 3 months
  Change in pocket depth between baseline and 3-month post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- National Obesity Centre, Yaoundé, Cameroon

REFERENCES:
- [Derived] Tsobgny-Tsague NF, Lontchi-Yimagou E, Nana ARN, Tankeu AT, Katte JC, Dehayem MY, Bengondo CM, Sobngwi E. Effects of nonsurgical periodontal treatment on glycated haemoglobin on type 2 diabetes patients (PARODIA 1 study): a randomized controlled trial in a sub-Saharan Africa population. BMC Oral Health. 2018 Feb 26;18(1):28. doi: 10.1186/s12903-018-0479-5. PMID 29482543